CLINICAL TRIAL: NCT04762121
Title: Preliminary Prospective Observational Study on Peripheral Intravenous Catheter Insertion
Brief Title: Observational Peripheral IV Insertion Study
Status: Withdrawn | Type: Observational
Why Stopped: Investigators left the institution
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: EX070
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Pain, Acute; Satisfaction
MeSH Terms: conditions — Acute Pain; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients requiring intravenous catheter insertion: Adults (>18 years old) who require intravenous catheter insertion for their operation/procedure
  Interventions: Procedure: Peripheral IV

INTERVENTIONS:
Procedure: Peripheral IV — Insertion of peripheral intravenous catheter

SUMMARY:
IV placement is a common and necessary for surgical procedures. Unfortunately, pain associated with needle catheterization experienced during peripheral IV placement is a source anxiety and discomfort in many patients. The intensity of pain and distress caused by procedures can vary from mild to moderate, but also may be severe in certain patients resulting in numerous physiological, psychological, and emotional consequences. As such, the investigators ultimately aim to evaluate the techniques that could make the placement of the IV more comfortable.

DETAILED DESCRIPTION:
As a preliminary study, the investigators are interested in conducting a prospective observational study to collect baseline data to characterize and collect baseline data on pain associated with needle catheterization in the hospital.

Many factors including size of needle, experience of the individual placing IV, previous history of depression may vary the IV placement experience of a patient; however, only some of these factors may directly affect the magnitude of pain experienced by a patient. Currently, there is limited literature available on what factors affect the pain/satisfaction patients experience with IV insertion. Soysal et al. have previously reported that depressed patients reported higher severity of pain during IV catheter placement than non-depressed patients in a cross-sectional, observational study (n= 925). The authors have also demonstrated that age, sex, site of IV catheter insertion, use of antidepressant drugs, and whether the individual placing the IV catheter is a nurse or physician do not affect the magnitude of pain. Similarly, Van Loon et al have demonstrated that insertion of a smaller sized peripheral intravenous catheter did not result in lower pain sensation. However, Galvin et al. conducted a randomized clinical trial that demonstrated that the site of IV catheter insertion makes a difference in the pain patients feel during IV catheter insertion. Furthermore, no study exists that has investigated whether patients experience a different magnitude of pain when different levels of physician trainees place the IV catheter. Also, no study exists that compares whether peripheral IV cannulation with no pain relief method versus intradermal lidocaine 1% injection versus intradermal lidocaine 2% injection versus Buzzy® device affect the pain/satisfaction that patients experience with IV catheter insertion.

Through the conduction of this study, the investigators hope to further evaluate which factors and techniques affect the experience patients have with peripheral IV cannulation; this knowledge could help the investigators figure out ways to make IV cannulation as comfortable as possible for patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18 to 99
* Patients requiring intravenous catheter insertion for their operation/procedure.

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients requiring intravenous catheter insertion for their operation/procedure.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-02-12 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Pain with IV Cannulation based on the Visual Analog Scale | 5-20 minutes
  How much pain do adult patients experience with peripheral IV cannulation with no pain relief method versus intradermal lidocaine 1% injection versus intradermal lidocaine 2% injection versus Buzzy® device? The Visual Analog Scale is used for linear measurement of pain, where the minimum number is 0 (no pain) and the maximum number is 10 (unimaginable pain).

SECONDARY OUTCOMES:
Satisfaction with IV cannulation based on the Numerical Rating Scale | 5-20 minutes
  How much satisfaction do adult patients experience with peripheral IV cannulation with no pain relief method versus intradermal lidocaine 1% injection versus intradermal lidocaine 2% injection versus Buzzy® device? The Numerical Rating Scale is used for linear measurement of satisfaction, where the minimum number is 1 (very dissatisfied) and the maximum number is 5 (very satisfied).
Pain related to IV location based on the Visual Analog Scale | 5-20 minutes
  Does location of the peripheral intravenous catheter placement affect the pain that adult patients experience with peripheral IV cannulation? The Visual Analog Scale is used for linear measurement of pain, where the minimum number is 0 (no pain) and the maximum number is 10 (unimaginable pain).
Pain related to IV size based on the Visual Analog Scale | 5-20 minutes
  Does size of the peripheral intravenous catheter affect the pain that adult patients experience with peripheral IV cannulation? The Visual Analog Scale is used for linear measurement of pain, where the minimum number is 0 (no pain) and the maximum number is 10 (unimaginable pain).
Pain from IV insertion related to stage of the training of the healthcare provider based on the Visual Analog Scale | 5-20 minutes
  Does the stage of the training of the healthcare provider affect the pain that adult patients experience with peripheral IV cannulation? The Visual Analog Scale is used for linear measurement of pain, where the minimum number is 0 (no pain) and the maximum number is 10 (unimaginable pain).
Pain from IV insertion based on the Visual Analog Scale related to history of patient having anxiety | 5-20 minutes
  Does the history of patient having anxiety affect the pain that adult patients experience with peripheral IV cannulation? The Visual Analog Scale is used for linear measurement of pain, where the minimum number is 0 (no pain) and the maximum number is 10 (unimaginable pain).
Pain from IV insertion based on the Visual Analog Scale related to history of patient having depression | 5-20 minutes
  Does the history of patient having depression affect the pain that adult patients experience with peripheral IV cannulation? The Visual Analog Scale is used for linear measurement of pain, where the minimum number is 0 (no pain) and the maximum number is 10 (unimaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- St. Elizabeth's Medical Center, Brighton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No